CLINICAL TRIAL: NCT00852488
Title: A Medium-term Venous Access Alternative in Infants Undergoing Congenital Heart Surgery
Brief Title: Medium-term Venous Access in Congenital Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Bichell, Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #080906
Record Dates: First submitted 2009-02-04; First posted 2009-02-27 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2010-02

CONDITIONS: Congenital Heart Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Catheter (Experimental): Cohort undergoing catheter placement using the new technique being studied
  Interventions: Procedure: Placement of transthoracic catheter

INTERVENTIONS:
Procedure: Placement of transthoracic catheter — Placement of transthoracic catheter into the inferior vena cava
  Other Names: Bard; transthoracic catheter

SUMMARY:
This study is designed to evaluate medium-term central venous catheter placement in infants undergoing complex cardiac surgery using a new technique. This technique involves placement of the catheter into the inferior vena cava through a subcutaneous tunnel and through a tunnel between pericardium and diaphragm.

ELIGIBILITY:
Inclusion Criteria:

* Infants undergoing surgical correction or palliation of congenital heart disease via sternotomy
* Age 0-365 days
* Anticipated intensive care stay over 10 days
* Need for central venous access or prolonged venous access

Exclusion Criteria:

* Presence of access that is likely to last more than 10 days at time of operation
* Septic shock
* Known inferior vena cava thrombosis
* Operations not approached by sternotomy

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Days of complication-free use. Morbidity (infection, malposition, bleeding, thrombosis, need for removal for catheter-related complication). Need for additional catheter placement or reintervention. | Until catheter no longer needed; it is not anticipated that these remain longer than 2 weeks. Prior to discharge all will have been removed and final assessment of primary outcome will be obtained

CONTACTS AND LOCATIONS:
Overall Officials: David P Bichell, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States